CLINICAL TRIAL: NCT05433181
Title: A Phase 1/2, Randomized Double-blind Placebo-Controlled Trial to Test the Safety and Antiviral Activity of ACE2 Chewing Gum on SARS-CoV-2 Viral Load (COVID 19)
Brief Title: ACE2 Chewing Gum on SARS-CoV-2 Viral Load (COVID 19)
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: For administrative reasons, the study was never opened and was terminated.
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 851459
Record Dates: First submitted 2022-06-24; First posted 2022-06-27 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: SARS-CoV-2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ACE2 Chewing Gum (Experimental)
  Interventions: Drug: ACE2 Chewing Gum
- Placebo Chewing Gum (Placebo Comparator)
  Interventions: Other: Placebo Chewing Gum

INTERVENTIONS:
Drug: ACE2 Chewing Gum — The IP is formulated as an oral plant powder, which is packaged into a chewing gum. No specific excipient, buffer, salt or pH is required. CTB-ACE2, with efficient binding to both GM1 and ACE2 receptors, effectively blocks binding of the spike protein and viral entry into human cells. Oral epithelial cells are enriched with both receptors. In addition, ACE2 directly binds to the spike protein and inactivates SARS-CoV-2 virus. Therefore, CTB-ACE2 chewing gum is being evaluated for impact on entry and transmission of SARS-CoV-2.
  Arms: ACE2 Chewing Gum
Other: Placebo Chewing Gum — Chewing gum containing wild-type lyophilized plant cells manufactured to match the IP.
  Arms: Placebo Chewing Gum

SUMMARY:
A randomized double-blind, placebo controlled clinical trial of the safety, tolerability, and antiviral activity of angiotensin-converting enzyme 2 (ACE2) chewing gum over a 3-day period in non-hospitalized subjects with Severe Acute Respiratory Syndrome Coronavirus 2 (SARS-CoV-2) infection.

ELIGIBILITY:
Inclusion Criteria:

1. Able and willing to provide informed consent prior to initiation of study procedures.
2. Stated willingness to comply with all study procedures and availability for the duration of the study.
3. Male or female, aged 18 years to 65 years.
4. Had a positive PCR or antigen test for SARS-CoV-2 within 72 hours of enrollment.
5. In the opinion of the investigator, has the ability to comply with study procedures including chewing the study products (gum).
6. Stated willingness to refrain from brushing, eating or using any oral health care products, including mouth rinses at least one hour prior to first saliva sample.
7. Stated willingness to abstain from eating mints or other chewing gums during the duration of the study.
8. Stated willingness to abstain from using mouth rinse/gargling solutions at the time of enrollment and for the duration of the study.
9. Stated willingness to use an acceptable method of birth control throughout duration of the study. Acceptable methods include hormonal contraceptives, barrier methods, abstinence, or other effective methods approved by the PI.
10. Stated ability and willingness to store saliva samples at approximately 40° F for 3 days.

Exclusion Criteria:

1. Individuals receiving antiviral medications that are thought to be active against SARS-CoV-2 in the opinion of the investigator.
2. Individuals receiving oral or injectable antimicrobial medications (antibacterial, antiviral, antibiotics, including hydroxychloroquine) at time of enrollment.
3. Currently undergoing cancer treatment.
4. Pregnant or breastfeeding women.
5. Participation in any other clinical trial within the past 14 days that used an investigational drug product.
6. Admitted to the hospital or other medical facility or in the opinion of the investigator expected to require admission to a medical facility for the duration of the study.
7. Taking chronic immunosuppressive medications at time of enrollment, defined as immunomodulatory agents or a prednisolone dose greater than 10 mg a day.
8. Uncontrolled hypertension, defined as ≥160 mmHg systolic or ≥100 mmHg diastolic.
9. Allergy/hypersensitivity to lettuce, gelatin (plant based), stevia, or unwillingness to consume genetically modified plant material.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-02 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Evaluate the safety and tolerability of CTB-ACE2 chewing gum. | At time of consent through Day 28
  The safety and tolerability in COVID 19+ adult individuals as measured by frequency of solicited adverse events (AEs).

SECONDARY OUTCOMES:
Test the antiviral activity of ACE2 chewing gum on reducing SARS-CoV-2 viral load in the oral cavity of COVID-19+ individuals via authorized PCR. | Days 1-4
  The change in amount of SARS-CoV-2 in saliva before and after intervention (chewing gum for 10 minutes) via authorized PCR; this includes after first use and sustained use over 3 days.
Evaluate the Symptom score of documented SARS-CoV-2 infection relative to treatment group (CTB-ACE2 chewing gum/placebo). | Days 1-4
  Symptom score of documented SARS-CoV-2 infection relative to treatment group (CTB-ACE2 chewing gum/placebo).

OTHER OUTCOMES:
Test the antiviral activity of ACE2 chewing gum on reducing SARS-CoV-2 viral load in the oral cavity of COVID-19+ individuals via antigen quantitation analysis. | Days 1-4
  The change in amount of SARS-CoV-2 in saliva before and after intervention (chewing gum for 10 minutes) via antigen quantitation analysis; this includes after first use and sustained use over 3 days.

CONTACTS AND LOCATIONS:
Locations (1):
- Infectious Diseases Clinical Trial Unit, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ganesan PK, Kulchar RJ, Kaznica P, Montoya-Lopez R, Green BJ, Streatfield SJ, Daniell H. Optimization of biomass and target protein yield for Phase III clinical trial to evaluate Angiotensin Converting Enzyme 2 expressed in lettuce chloroplasts to reduce SARS-CoV-2 infection and transmission. Plant Biotechnol J. 2023 Feb;21(2):244-246. doi: 10.1111/pbi.13954. Epub 2022 Dec 1. No abstract available. PMID 36314106